CLINICAL TRIAL: NCT00492661
Title: A Pilot Trial of the Effect of Dietary and Exercise Intervention on Insulin Resistance and Metabolic Parameters in De Novo Renal Transplant Recipients on Prograf (Tacrolimus)
Brief Title: A Pilot Trial to Evaluate the Effect of Diet and Exercise in Renal Transplant Recipients on Tacrolimus
Acronym: PRIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR013702; OTH/506TRA4004
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Renal Transplantion; Kidney Transplantion
Keywords: Tacrolimus; Prograf; PRIDE
MeSH Terms: interventions — Tacrolimus; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus With Diet and Exercise Intervention (Experimental): Participants on tacrolimus for immunosuppression (drug which suppresses the body's immune response, used in transplantation and diseases caused by disordered immunity) will be provided with intensive dietary advice and supervised progressive resistance training (PRT) for a period of 6 months. Dosage and administration of tacrolimus will be as per Investigator's discretion.
  Interventions: Drug: Tacrolimus With Diet and Exercise Intervention

INTERVENTIONS:
Drug: Tacrolimus With Diet and Exercise Intervention — Participants on tacrolimus for immunosuppression will be provided with intensive dietary advice and supervised for a period of 6 months. Dosage and administration of tacrolimus will be as per Investigator's discretion.
  Other Names: Prograf

SUMMARY:
The purpose of this trial is to investigate whether a combined dietary and exercise intervention, added to standard care, reduces the expected frequency of insulin resistance in renal (kidney) transplant recipients on tacrolimus.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (study following participants forward in time), single-arm, multi-center (conducted in more than 1 center), interventional pilot study of the effects of a combined dietary and exercise intervention on glucose metabolism. The duration of this study will be 6 months and will include following visits: Baseline, Week 4, Week 12, and Week 24. Dietary compliance will be evaluated with a 3-day food record and during weekly telephone conversations and face-to-face visits with a dietician. Exercise compliance will be measured using an exercise log presented to the co-ordinator at the end of each month. Primarily, participants with insulin resistance will be assessed by Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) of greater than 1 at 6 months. Participants' safety and tolerability will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who has sufficiently recovered from surgery to tolerate an intensive exercise evaluation
* Participants who have received a living-donor or cadaveric (from dead donor) renal transplant
* Participants who has been initiated tacrolimus as first-line immunosuppressive agent
* Participants who has given informed consent forms

Exclusion Criteria:

* Participants with significant disease or disability that prevents taking part in a diet or exercise regime (e.g. cardiac instability, including unstable angina [chest pain due to decreased oxygen being supplied to the heart] and/or other unstable disease, severe cognitive [mental functioning] impairment)
* Participants with significant post-surgical complications that prevent participation in the exercise component of the study (e.g. wound dehiscence [pathologic process consisting of a partial or complete disruption of the layers of a surgical wound] or infection)
* Participants with contraindications to maximal exercise testing or high-intensity progressive resistance training (e.g. proliferative diabetic or hypertensive retinopathy, un-repaired aneurysm, critical aortic stenosis, recurrent symptomatic hernias, New York Heart Association (NYHA) class-IV congestive heart failure)
* Participants with non-ambulatory (mobility) status
* Participants who require ongoing systemic immunosuppressive therapy for an indication other than renal transplant and this therapy is higher than that required for their kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Insulin Resistance | Week 24
  Percentage of participants with insulin resistance as defined by a Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) greater than 1. HOMA uses fasting glucose and insulin (or C-peptide) to assess beta-cell function and IR. HOMA-IR is used to estimate insulin resistance. HOMA-IR is calculated by equation: HOMA-IR=fasting plasma insulin (milliunit [mU] per liter [L]) * fasting plasma glucose (millimole per liter [mmol per L]) divided by 22.5.

SECONDARY OUTCOMES:
Percentage of Participants With Impaired Fasting Glycaemia (IFG) | Week 24
  IFG is defined as a fasting venous plasma glucose concentration greater than or equal to 6.1 mmol per L but less than 7.0 mmol per L, together with a 2-hour plasma glucose concentration of less than 7.8 mmol per L.
Percentage of Participants With Impaired Glucose Tolerance (IGT) | Week 24
  IGT is defined as fasting venous plasma glucose of less than 7.0 mmol per L, together with a 2-hour plasma glucose of greater than or equal to 7.8 mmol per L but less than 11.1 mmol per L.
Percentage of Participants With Diabetes Mellitus (DM) | Week 24
  DM is defined as a fasting plasma glucose concentration greater than or equal to 7.0 mmol per L, or a 2-hour plasma glucose greater than or equal to 11.1 mmol per L.
Beta Cell Function | Baseline, Week 4, Week 12, and Week 24
  HOMA-Beta is used to assess beta-cell function. HOMA-Beta is a measure of Beta-cell function (higher values present increased insulin secretion for a given glucose level). HOMA-Beta is calculated by the equation: HOMA-Beta=(20*FPI) divided by (FPG-3.5), where, FPI is fasting plasma insulin concentration (mU per L) and FPG is fasting plasma glucose concentration (mmol per L).
Number of Participants With Acute Rejection, Graft Loss and Death | Week 24
  Acute rejection episodes are classified into: Spontaneously resolving - a rejection episode which is not treated with new or increased corticosteroid medication, antibodies or any other medication. Corticosteroid sensitive - a rejection episode, which is treated with new or increased corticosteroid medication only. Corticosteroid resistant - a rejection episode, which is not resolve following treatment with corticosteroids. Graft loss is defined as re-transplantation, nephrectomy, death or as dialysis ongoing at study end (or at withdrawal of the participants from the study).
Body Mass Index (BMI) | Baseline, Week 4, Week 12 and Week 24
  BMI is a statistical measurement which compares a person's weight and height. Though it does not actually measure the percentage of body fat, it is used to estimate a healthy body weight based on participant's height. BMI is equal to weight divided by height square. Weight is measured in Kilogram and height is measured in meter.
Bone Mineral Density | Baseline and Week 24
  Bone mineral density is measured by Dual-Energy X-ray Absorptiometry (DEXA).
Waist to Hip Ratio (WHR) | Baseline, Week 4, Week 12 and Week 24
  WHR is performed using a standard medical measuring tape, with recordings documented in centimeters. Measurements will be compared against data from participating sites (where available) and against baseline. Measurement of hip circumference will be performed at the widest part of the buttocks. Measurement of the waist will be performed at the smaller circumference of the natural waist (usually just superior to the umbilicus). WHR is calculated by dividing the waist measurement by the hip measurement, and recorded to 2 decimal places.
Body Composition: Percent Body Fat | Baseline and Week 24
  Body fat will be assessed by DEXA scan.
Body Composition: Lean Mass, Bone Mass and Adjusted Weight | Baseline and Week 24
  Body composition lean mass and bone mass will be assessed by DEXA scan.
Body Composition: T Score (Full Body) and Z Score (Full Body) | Baseline and Week 24
  Body composition: T score (Full body) and Z score (full body) will be assessed by DEXA scan.
Blood Pressure: Systolic and Diastolic Pressure | Baseline, Week 4, Week 12 and Week 24
  Measurement of blood pressure will be performed by using a completely automated device consisting of an inflatable cuff and oscillatory detection system. Blood pressure will be taken supine, after 5 minutes of rest.
Lipid Profile | Baseline, Week 4, Week 12, and Week 24
  In lipid profile total cholesterol, high-density lipoprotein (HDL) - cholesterol, low-density lipoprotein (LDL) - cholesterol and triglycerides levels will be evaluated. Measurement of the lipid profile will be performed in fasted state.
Hemoglobin A, Glycosylated (HbA1c) | Baseline, Week 4, Week 12 and Week 24
  Measurement of the change in HbA1c will be performed in fasted state and in local laboratories.
Estimated Glomerular Filtration Rate (eGFR) | Baseline, Week 4, Week 12 and Week 24
  The eGFR is calculated by Modification of Diet in Renal Disease (MDRD) equation is recommended by Kidney Health Australia as the calculation of choice for predicting GFR. According to MDRD equation eGFR is equal to 186*(Serum creatinine/0.095)^-1.154*age^0.203*race*sex, where the unit of serum creatinine is micro mole per L, the age is in years; race is 1.212 if African American, or 1 otherwise; and sex equals 1 if male, and 0.742 if female. eGFR will be compared against baseline.
36-Item Short-Form (SF-36) Score - Health Survey | Baseline, Week 12 and Week 24
  This SF-36 standardize survey evaluates participants health by 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as Physical Component Scores (PCS) and Mental Component Scores (MCS). The score for a section is an average of the individual question scores, which are scaled 0 to 100, Higher score indicates highest level of functioning.
Percentage of Participants who will be Sedentary, Insufficiently Active and Sufficiently Active According to Active Australia Survey (AAS) | Week 4, Week 12 and Week 24
  AAS is used for physical activity surveillance and it consists of following categories: 'sedentary' - people who are doing no activity at all; 'sufficiently active'- participation in at least 150 minutes per week; 'insufficiently active'- the remainder participants whose participation is not enough to obtain a health benefit.
Percentage of Participants Compliant With Both Dietary Advice and Exercise Program and Non-Compliant With Dietary Advice or Exercise Program | Week 4, Week 12 and Week 24
  Compliance with dietary advice will be measured on a categorical scale ranging from 0=no compliance to 10=full compliance. Compliance with exercise program is measured as the completion of 3 exercise sessions per week for the 6-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd
Locations (4):
- Australia (4):
  - Camperdown
  - Clayton
  - Perth
  - Woodville

REFERENCES:
- See also: A Pilot Trial of the Effect of Dietary and Exercise Intervention on Insulin Resistance and Metabolic Parameters in De Novo Renal Transplant Recipients on Prograf (Tacrolimus) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=237&filename=CR013702_CSR.pdf